CLINICAL TRIAL: NCT03524352
Title: Prospective Multicenter Randomized Controlled Double-blind Label Study of the Prophylaxis of Recurrent Pouchitis After Fecal Microbiota Transplant in UC With Ileo-anal Anastomosis
Brief Title: the Prophylaxis of Recurrent Pouchitis After Fecal Microbiota Transplant in UC With Ileo-anal Anastomosis
Acronym: POCA
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RC17_0021
Record Dates: First submitted 2018-05-02; First posted 2018-05-14 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Pouchitis
Keywords: recurrent pouchitis; fecal microbiota transplant
MeSH Terms: conditions — Pouchitis | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- fecal microbiota (Experimental)
  Interventions: Other: fecal microbiota
- placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Other: fecal microbiota — fecal microbiota in suspension
  Arms: fecal microbiota
Other: Placebo — sterile saline
  Arms: placebo

SUMMARY:
Ulcerative colitis (UC) is a chronic inflammatory digestive (IBD) disease medically treated with corticosteroids, aminosalicylates, immunomodulators, and biologics. Almost one third of UC patients will require surgical interventions because of fulminant colitis, dysplasia, cancer, or medical refractory diseases. Restorative proctocolectomy with ileal pouch-anal anastomosis (IPAA) is the current standard surgical intervention. Anastomotic leak, pouch failure, pelvic sepsis, and pouch ischemia can occur after the procedure, but the most common long-term complication is pouchitis, an idiopathic inflammatory condition involving the ileal reservoir. Symptoms of pouchitis are increased stool frequency, urgency, incontinence, bloody stools, abdominal or pelvic discomfort, fatigue, malaise, and fever. The prevalence of pouchitis ranges from 23 to 46 %, with an annual incidence up to 40 %. Though the majority of initial cases of pouchitis are easily managed with a short course of antibiotics, in about 5 to 15 % of cases, inflammation of the pouch becomes chronic with very few treatments available.

Fecal microbiota transplantation (FMT) is a novel therapy to transfer normal intestinal flora from a healthy donor to a patient with a medical condition potentially caused by disrupted homeostasis of intestinal microbiota or dysbiosis. FMT has been widely used in refractory Clostridium difficile infection (CDI) and recently it has gained popularity for treatment of inflammatory bowel disease (IBD). Previous studies suggested that manipulating the composition of intestinal flora through antibiotics, probiotics, and prebiotic achieved significant results for treating acute episodes of UC-associated pouchitis. However, currently there is no established effective treatment for chronic antibiotic dependent pouchitis. Our project aims to evaluate the delay of relapse in chronic recurrent pouchitis after FMT versus sham transplantation.

ELIGIBILITY:
4.2. INCLUSION CRITERIA

Subjects must satisfy the following criteria to be enrolled in the study:

1. Male or female ≥ 18 years at the time of signing the informed consent form (ICF).
2. Subject must understand and voluntarily sign an ICF prior to conduct the study related assessments/procedure.
3. Willing and able to adhere to the study visit scheduled and other protocol requirements.
4. Subjects must have been operated with ileal pouch anal anastomosis (IPAA) with a duration of at least 6 month prior the screening visit.
5. Subject must have a diagnosis of recurrent pouchitis defined as at least 2 episodes in the last year or relapsing immediately after a reasonable response to antibiotherapy (the antifungal medication is allowed until the day before transplantation).
6. Subject must be in remission with a Pouchitis Disease Activity Index (PDAI) < 7 at the screening
7. Subject must affiliation with social security system or beneficiary from such system
8. Female of childbearing potential must have a negative pregnancy test at screening and must agree to practice effective methods of contraception

4.3. NON-INCLUSION CRITERIA

Subjects who meet any of the following non inclusion criteria could not be enrolled in this study:

1. Crohn disease or indeterminate colitis
2. Anastomotic stenosis
3. Subject with prior treatment by probiotic within 3 month prior to the transplantation visit
4. Subject with prior treatment by corticosteroids within 6 weeks prior to the transplantation visit
5. Subject with prior treatment by immunosuppressors within 3 month prior to the transplantation visit unless treatment has been introduced for more than 8 weeks at a stable dose.
6. Prior treatment with a biologic within 3 month prior the transplantation visit unless treatment has been introduced for more than 8 weeks at a stable dose.
7. Documented active infection of any kind in the last 6 months likely to require anti-infective treatment during the next months
8. Absolute neutrophil count (ANC) < 1.5 x 109 /L (1,500 mm3)
9. Infection with chronic HIV
10. Pregnant female or breastfeeding
11. Chronic medical or psychiatric disease that may interfere with subject's ability to comply with study procedures
12. Administration of investigational drug within 3 months prior to planned FMT
13. Adults under guardianship, Safeguard justice or trusteeship
14. Subject with difficulty in follow-up (vacation, job transfer, geographical distance, lack of motivation).
15. Patients with contraindication to colonoscopy or anesthesia (if necessary)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2020-03-12 (Actual); Primary Completion 2028-05-12 (Estimated); Study Completion 2028-05-12 (Estimated)

PRIMARY OUTCOMES:
Number of days between the date of transplantation and the date of relapse according to physiological and endoscopic parameter (pochitis disease activity index) | 106 weeks

SECONDARY OUTCOMES:
Number of relapse rate according to physiological and endoscopic parameter (pochitis disease activity index) | 24 weeks
Number of relapse rate according to pochitis disease activity index (physiological and endoscopic parameter) | 52 weeks
Number of days within the transplantation and the instauration of an antibiotherapy or alternative treatment | 52 weeks
Number of adverse events | 104 weeks
Number of fecal microbiota engraftment by 16S sequencing | 8 weeks
Number of evolution of health-related to disability according to physiological and endoscopic parameter (pochitis disease activity index) | weeks -5
Number of evolution of health-related to disability according to physiological and endoscopic parameter (pochitis disease activity index) | 0 week
Number of evolution of health-related to disability according to physiological and endoscopic parameter (pochitis disease activity index) | 8 weeks
Number of evolution of health-related to disability according to physiological and endoscopic parameter (pochitis disease activity index) | 24 weeks
Number of evolution of health-related to disability according to physiological and endoscopic parameter (pochitis disease activity index) | 52 weeks

CONTACTS AND LOCATIONS:
Locations (13):
- France (13):
  - CHU Angers, Angers
  - CHU Estaing, Clermont-Ferrand
  - Hopital Beaujon, Clichy, Clichy
  - CHU Henry Mondor, Créteil
  - CHU Claude Huriez, Lille
  - CHU Lyon Sud, Lyon
  - CHRU Nancy, Nancy
  - CHU of Nantes, Nantes
  - CHU de l'Archet 2, Nice
  - Hopital Saint Antoine, Paris
  - Groupe Hospitalier Sud- Hopital Haut-lévêque, Pessac
  - CHU Pontchaillou, Rennes
  - CHU Toulouse, Toulouse

REFERENCES:
- [Derived] Trang-Poisson C, Kerdreux E, Poinas A, Planche L, Sokol H, Bemer P, Cabanas K, Hivernaud E, Biron L, Flet L, Montassier E, Le Garcasson G, Chiffoleau A, Jobert A, Lepelletier D, Caillon J, Le Pape P, Imbert BM, Bourreille A. Impact of fecal microbiota transplantation on chronic recurrent pouchitis in ulcerative colitis with ileo-anal anastomosis: study protocol for a prospective, multicenter, double-blind, randomized, controlled trial. Trials. 2020 Jun 3;21(1):455. doi: 10.1186/s13063-020-04330-1. PMID 32493442